CLINICAL TRIAL: NCT02804984
Title: Identification of Molecular Defects in Idiopathic Cytopenia of Undetermined Significance
Acronym: AMICUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2014_843_0008
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Myelodysplastic Syndromes
Keywords: idiopathic cytopenia of undetermined significance (ICUS); molecular defects
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * blood
  * bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICUS: idiopathic cytopenia of undetermined significance (ICUS)
  Interventions: Genetic: ICUS

INTERVENTIONS:
Genetic: ICUS

SUMMARY:
The project's objective is to identify and characterize somatic mutations in cases of idiopathic cytopenia of undetermined significance (ICUS) on the basis of molecular defects found in myelodysplastic syndrome (MDS), in order to validate the hypothesis whereby ICUS may be a precursor of MDS

DETAILED DESCRIPTION:
The project's objective is to identify and characterize somatic mutations in cases of idiopathic cytopenia of undetermined significance (ICUS) on the basis of molecular defects found in myelodysplastic syndrome (MDS), in order to validate the hypothesis whereby ICUS may be a precursor of MDS. To this end, high-throughput exon sequencing (using next-generation sequencing (NGS)) will be used to target the genes known to be mutated in MDS. This study is important for two reasons. Firstly, it will help to optimise the clinical monitoring of patients with molecular defects and considered to be at risk of progression. Secondly, it will provide a better understanding of the fundamental molecular mechanisms underlying the progression of ICUS to MDS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over.
* Haemoglobin <11 g/dl and/or a polynuclear neutrophil count <1.5.109/L and/or a platelet count <100.109/L
* Full clinical biochemistry/haematological profiling: complete blood count, blood smear, reticulocyte count, iron status, folates, B12, TSH, creatinine, liver enzymes, ANAs, rheumatoid factor, anticardiolipin antibodies, Coombs test, EPO assay, serological tests for HIV, HVB and HVC.
* Availability of a bone marrow differential cell count and an evaluation of myelopoiesis disorders (number of lineages, percentage of cells affected, etc.) plus Perls staining.
* Availability of a cytogenetic analysis.
* Voluntary provision of written, informed consent
* Life expectancy >6 months
* Social security coverage

Exclusion Criteria:

* An obvious cause of anaemia (if isolated): iron deficiency, chronic kidney failure (clearance <60 ml/min), regenerative anaemia (reticulocytes >150G/L)
* Vitamin B12 or B9 deficiency
* Hepatomegaly, or clinical and/or ultrasound signs of portal hypertension
* Clinical and/or ultrasound signs of splenomegaly
* Abnormal liver enzyme levels: total bilirubin, alkaline phosphatases or transaminases > 1.5N; gammaGT > 2N. A history of (or diagnostic criteria during screening) auto-immune diseases such as systemic erythematous lupus, antiphospholipid syndrome or Evans syndrome.
* An abnormal bone marrow differential cell count
* A bone marrow karyotype revealing MDS
* Medical, psychological or social conditions that prevent the participant from correctly understanding the study procedures.
* Legal guardianship and incarceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with myelodysplastic syndrome
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
high-throughput sequencing | Day 0
  The presence or absence of one or several of the following molecular defects, as detected by high-throughput sequencing: DNMT3A, TET2, IDH1/2, ASXL1, EZH2, RUNX1, EVI1, GATA2, P53, JAK2, CBL, KRAS, SF3B1, SRSF2, U2AF1, and ZRSR2.

SECONDARY OUTCOMES:
phenotypic defects | Day 0
  Analysis of phenotypic defects detected by flow cytometry.
growth of erythroid progenitors | Day 0
  Analysis of the growth of erythroid progenitors (BFU-E) and granulocyte-monocyte progenitors (CFU-GM).
Appearance of MDS | 6 months
  Appearance of MDS during follow-up: a bone marrow differential cell count at 6 months and whenever cytopenia appears.

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère GRUSON, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France